CLINICAL TRIAL: NCT05245383
Title: Skin Irritation Test of Ten Products
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 202107020RSD
Record Dates: First submitted 2021-12-23; First posted 2022-02-17 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-11

CONDITIONS: Dermatitic Reaction of Face
Keywords: skin; skin health; allergen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other)
  Interventions: Other: ten products (S01~S10) and two blank (BK1, BK2)

INTERVENTIONS:
Other: ten products (S01~S10) and two blank (BK1, BK2) — S01 "Functional Peptides Recovering Essence EX" S02 "Advanced Revitalizing Eye Cream" S03 "Advanced Revitalizing Lotion" S04 "NB-1 Anti-Sensitive Repair Activator" S05 "NB-1 Anti-Sensitive Repair Toning Extract" S06 "Ginseng Vitality Serum" S07 "Ginseng Revitalizing Age-defense Essence Cream" S08 "Ginseng Age-defense Eye Cream" S09 "Revital Energy Balance Gel" S10 "Revital Energy Tightening Body Lotion" BK1 "Water" BK2 "Blank" ten products and two blank, 24 hours single application patch test on the back.

SUMMARY:
Evaluation of cutaneous tolerance of ten products by primary irritant patch test

DETAILED DESCRIPTION:
The purpose of this clinical study was the evaluation of skin irritation potential of ten products after a single application under occlusive patch on human skin.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 70 years old, healthy male and female (sex ratio 1:1)
* No acute or chronic diseases including skin diseases.
* No current medications.

Exclusion Criteria:

* Pregnancy or breast feeding.
* Abnormal blood test result/results (evaluation criteria: WBC, AST, ALT, and Creatinine)
* Back skin with moles, acne, tattoo, scars, red spots, burns, etc.
* Current dermatology medication which might affect skin condition evaluation.
* Current irritated reaction on test site.
* Participating in other clinical trial(s) within 7 days.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-04-29 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety/Adverse Event Outcome Measure | Up to 48 hours
  Number of participants with Serous and Non-Serous Adverse Event
Total Number of Positive Responses Across All Participants | Reading results at 30 minutes, 24 hours and 48 hours after the removal of the test products.
  Change from baseline of test products by using ICDRG (International Contact Dermatitis Research Group) grading

CONTACTS AND LOCATIONS:
Overall Officials: SUNG-JAN LIN, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horita K, Tanoue C, Yasoshima M, Ohtani T, Matsunaga K. Study of the usefulness of patch testing and use test to predict the safety of commercial topical drugs. J Dermatol. 2014 Jun;41(6):505-13. doi: 10.1111/1346-8138.12505. PMID 24909212
- [Background] Fullerton A, Benfeldt E, Petersen JR, Jensen SB, Serup J. The calcipotriol dose-irritation relationship: 48 hour occlusive testing in healthy volunteers using Finn Chambers. Br J Dermatol. 1998 Feb;138(2):259-65. doi: 10.1046/j.1365-2133.1998.02071.x. PMID 9602871